CLINICAL TRIAL: NCT00388453
Title: ADHERE Study: Application of Dx-pH Catheter for Extra-esophageal Reflux Evaluation
Brief Title: Efficacy of Dx-pH Probe in Diagnosing Extra-esophageal Reflux Disease
Acronym: ADHERE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigatori, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 060860
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: GERD; Larynx Disease
Keywords: Healthy volunteers
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngeal Diseases | interventions — Manometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Healthy volunteers with no history of GERD or EERD or Proton Pump Inhibitor (PPI) use
  Interventions: Device: Dx-pH Probe; Procedure: Manometry
- 2 (Experimental): subject is known to have GERD based on symptoms and previous positive response to PPI
  Interventions: Device: Dx-pH Probe; Procedure: Manometry
- 3 (Experimental): subject is known to have EERD based on symptoms and previous positive response to PPI
  Interventions: Device: Dx-pH Probe; Procedure: Manometry

INTERVENTIONS:
Device: Dx-pH Probe — 24 hour ph monitoring
Procedure: Manometry — procedure to measure pH at the Lower esophageal sphincter (LES) and Upper esophageal sphincter (UES)

SUMMARY:
The purpose of this study is to establish the clinical application of a new device that records pH changes in the hypopharynx. The investigators also aim to compare the consistency of distal esophageal pH with hypopharyngeal pH using both the "short" and the "long" catheters in patients.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) has been linked to many disorders and can be diagnosed through a variety of modalities utilizing 24 hour ambulatory pH monitoring which can register the duration, pattern and symptom correlation of distal esophageal acid exposure. This can be accomplished via a catheter probe connected from outside the body and placed through a nostril, advanced past the hypopharynx and down into the distal esophagus. Or, a small pH detector temporarily implanted in the distal esophagus during endoscopy can record reflux events. However, despite available technologies, there has long been a deficiency in detecting extra-esophageal reflux in the upper esophagus/ hypopharynx. This is of interest for gastroenterologists, otolaryngologists, and pulmonologists in the evaluation of extra-esophageal reflux as a potential culprit for asthma, chronic cough, laryngitis, globus, and non-cardiac chest pain. Until now, there has not been a device sensitive enough for accurately detecting extra-esophageal reflux (EERD) and clinicians have relied upon subjective response to empiric treatment with acid reducing medications to determine whether acid reflux was at the root of the symptoms. There are currently no well designed published studies with this device to assess its role in this group of difficult to treat patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers aged 18 to 65 years old.
2. Control group: No known history of GERD or EERD or prior PPI use.
3. GERD group: Patients with known history of GERD based on prior response to either histamine inhibitors (H2 blockers) or proton pump inhibitors (PPIs) and/or endoscopic esophagitis identified at endoscopy.
4. EERD group: Patients with chronic cough, asthma and laryngeal findings felt to be GERD related.

Exclusion Criteria:

1. Use of H2 blockers or PPIs within one week prior to and during the study for the GERD and EERD patients. No prior PPI use is allowed for the control population.
2. Use of antacids (Rolaids, Tums, Pepto-Bismol, etc.) within one day prior to or during the study.
3. Esophageal motility abnormalities (achalasia, esophageal spasm, severe dysphagia)
4. Expected non-compliance.
5. Positive history of ongoing alcohol or tobacco use and inability to refrain from using either during study duration (24 hours).
6. Recent nasal surgery or nasal obstruction.
7. Significant medical conditions that, in the investigator's judgment, would compromise the subject's health and safety (mental disability, psychiatric impairment, inability to read or comprehend the consent form)
8. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-10; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD, PhD, MS, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers for all three groups were recruited from the Vanderbilt Medical Center
Groups:
- Healthy Volunteers With no History of GERD or EERD or PPI Use: Healthy volunteers with no history of GERD or EERD or PPI use
  Dx-pH Probe: 24 hour ph monitoring
  Manometry: procedure to measure LES and UES
- Volunteers With History of Gastroesophageal Reflux Disease: Patients with a history of GERD symptoms (heartburn and/or regurgitation) at least once in a week in the past month and had an improvement of their symptoms with PPI use and if they had erosive esophagitis by Los Angeles classification at endoscopy.
- Volunteers With Laryngopharangeal Reflux (LPR): Patients suspected to have reflux-related laryngeal symptoms, including chronic cough, throat clearing and hoarseness. This group included non-smokers with unremarkable chest radiographs who had undergone extensive testing and exclusion of other common causes for their laryngeal symptoms by the Vanderbilt Allergy, Sinus and Asthma Program (ASAP), and Vanderbilt Voice Center (spirometry, methacholine challenge, sputum eosinophil count, otolaryngology exam, high-resolution computerized tomography scan of the thorax and sinuses and sinus testing).
Period: Overall Study
Arm/Group | Healthy Volunteers With no History of GERD or EERD or PPI Use | Volunteers With History of Gastroesophageal Reflux Disease | Volunteers With Laryngopharangeal Reflux (LPR)
Started | 20 | 17 | 10
Completed | 20 | 17 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Male and female normal volunteers who had no LPR symptoms or known history of GERD.
Groups:
- Volunteers With Gastroesophageal Reflux Disaese (GERD): History of GERD symptoms (heartburn and/or regurgitation) at least once in a week in the past month and had an improvement of symptoms with PPI use and if they had erosive esophagitis by LA classification at endoscopy
- Volunteers With Laryngopharangeal Reflux (LPR): Suspected to have reflux-related laryngeal symptoms, including chronic cough, throat clearing,and hoarseness.
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers With no History of GERD or EERD or PPI Use | Volunteers With Gastroesophageal Reflux Disaese (GERD) | Volunteers With Laryngopharangeal Reflux (LPR) | Total
Number analyzed (Participants) | 20 | 17 | 10 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 9 | 46
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 6 | 29
  Male | 8 | 6 | 4 | 18
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 10 | 47

OUTCOME MEASURES:

1. Primary Outcome: Decrease in pH From Baseline to <4
Description: The three study groups underwent dual pH measurements of the oropharyngeal as well as esophageal acid exposure employing the regular length probe for the oropharynx and the custom-designed long probe for the distal esophagus. The reason for the custom-designed esophageal measurement was to ensure that events noted in the oropharynx originated distally and were of gastric source. Measurements for the two locations were time synchronized to ensure accuracy. Calculations were based on length of time spent in upright and supine positions, and a combination of the two positions.
Time Frame: 24 hours
Population: Calculations were based on length of time spent in upright and supine positions, and a combination of the two positions.
Measure: Median (Inter-Quartile Range); unit: distal esophagus total % time pH <4
Groups:
- Volunteers With History of Gastroesophageal Reflux Disease: GERD symptoms (heartburn and/or regurgitation) at least once in a week in the past month with an improvement of symptoms with PPI use and if they had erosive esophagitis by LA classification at endoscopy.
- Volunteers With Laryngopharangeal Reflux (LPR): Suspected to have reflux-related laryngeal symptoms including chronic cough and hoarseness.
Arm/Group | Healthy Volunteers With no History of GERD or EERD or PPI Use | Volunteers With History of Gastroesophageal Reflux Disease | Volunteers With Laryngopharangeal Reflux (LPR)
Number analyzed (Participants) | 20 | 17 | 10
distal esophagus total % time pH <4 | 1.1 [0.5 to 3.9] | 3.2 [1.5 to 8.7] | 3.8 [1.8 to 6.7]
Statistical Analysis 1: Comparison: Healthy Volunteers With no History of GERD or EERD or PPI Use vs Volunteers With History of Gastroesophageal Reflux Disease vs Volunteers With Laryngopharangeal Reflux (LPR); Test type: Superiority or Other; p = .05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Decrease in pH From Baseline to <5
Description: The three study groups underwent dual pH measurements of the oropharyngeal as well as esophageal acid exposure employing the regular length probe for the oropharynx and the custom-designed long probe for the distal esophagus. The reason for the custom-designed esophageal measurement was to ensure that events noted in the oropharynx originated distally and were of gastric source. Measurements for the two locations were time synchronized to ensure accuracy. Calculations were based on length of time spent in upright and supine positions, and a combination of the two positions. Reflux event was calculated for a drop in pH from baseline to either <4, or <5, or <6 and each event had to last more than 5 seconds and could not be during the meals.
Time Frame: 24 hours
Population: Calculations were based on length of time spent in upright and supine positions, and a combination of the two positions. Reflux event was calculated for a drop in pH from baseline to either <4, or <5, or <6 and each event had to last more than 5 seconds and could not be during the meals.
Measure: Median (Inter-Quartile Range); unit: distal esophagus total % time pH <5
Arm/Group | Healthy Volunteers With no History of GERD or EERD or PPI Use | Volunteers With History of Gastroesophageal Reflux Disease | Volunteers With Laryngopharangeal Reflux (LPR)
Number analyzed (Participants) | 20 | 17 | 10
distal esophagus total % time pH <5 | 3.0 [1.9 to 8.3] | 6.5 [4.4 to 27] | 13 [3.6 to 19]

3. Primary Outcome: Decrease in pH From Baseline to <6
Description: as for outcome 2
Time Frame: 24 hours
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: distal esophagus total % time pH <6
Arm/Group | Healthy Volunteers With no History of GERD or EERD or PPI Use | Volunteers With History of Gastroesophageal Reflux Disease | Volunteers With Laryngopharangeal Reflux (LPR)
Number analyzed (Participants) | 20 | 17 | 10
distal esophagus total % time pH <6 | 11 [8.6 to 27] | 29 [12 to 54] | 31 [19 to 58]

4. Secondary Outcome: Number of Reflux Events
Description: Reflux event was calculated for a drop in pH from baseline to <6 and each event had to last more than 5 seconds and could not be during the meals.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: reflux events
Arm/Group | Healthy Volunteers With no History of GERD or EERD or PPI Use | Volunteers With History of Gastroesophageal Reflux Disease | Volunteers With Laryngopharangeal Reflux (LPR)
Number analyzed (Participants) | 20 | 17 | 10
reflux events | 6.5 [0.0 to 35] | 102 [5.0 to 181] | 75 [45 to 177]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Volunteers With Gastroesphageal Reflux Disease (GERD): GERD symptoms (heartburn and/or regurgitation) at least once in a week in the past month and an improvement of symptoms with PPI use and if they had erosive esophagitis by LA classification at time of endoscopy.
Arm/Group | Healthy Volunteers With no History of GERD or EERD or PPI Use | Volunteers With Gastroesphageal Reflux Disease (GERD) | Volunteers With Laryngopharangeal Reflux (LPR)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/10
Other Adverse Events (participants affected / at risk) | 1/20 | 0/17 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers With no History of GERD or EERD or PPI Use (N=20) | Volunteers With Gastroesphageal Reflux Disease (GERD) (N=17) | Volunteers With Laryngopharangeal Reflux (LPR) (N=10)
Cough (Gastrointestinal disorders) | 1 (1) | 0 | 0 — One patient reported a single episode of cough during the study.

LIMITATIONS AND CAVEATS:
Lack of prior validation studies on appropriate positioning of the oropharyngeal pH probe.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No